CLINICAL TRIAL: NCT03105830
Title: Pain Management Efficiency at Latent Period of Labour
Brief Title: Pain Management at Latent Period of Labour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Oleg Shnaider, head of delivery room, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0037-16-NHR-shnaider
Record Dates: First submitted 2017-02-06; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Labour
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention and data collection (Experimental): pain management by iv paracetamol
  Interventions: Drug: iv paracetamol

INTERVENTIONS:
Drug: iv paracetamol — iv paracetamol
  Other Names: perfalgan

SUMMARY:
Examine the effectiveness of an analgesic in PERFALGAN maternity latent phase of labor.

Examine the safety in PERFALGAN in the mother and the newborn in terms of the level of drug in blood

DETAILED DESCRIPTION:
Maternity are latent or first stage of labor and complained of pain at the level of 4 or higher on a scale VAS, and are not in risk (HIGH RISK). And did not receive analgesics within 4 hours.

The sample will consist of at least 100 women in labor.

1. women, will be identified in the reception room of a delivery room by midwives.
2. The research team will ask for consent after receiving an explanation and confirmation of understanding.
3. The midwife will perform and will record pain assessment by visual analog scores .
4. Maternity reported pain level 4 and above will be asked four questions out of data collection and offered them treatment I.V. PARACETAMOL 1gr as directed by the physician.
5. After giving I.V. PARACETAMOL 1g, carried out and documented estimate of the pain returns (by visual analog scores) after an hour wait at any time to wait four hours and two hours after birth.

   In cases of an outbreak of pain can give one of the following:

   Option A:

   Another portion of the I.V. PARACETAMOL 1gr within 4-6 hours the previous dose. The maximum daily dose of 4 grams.

   Option B:

   N2O by procedure

   A third possibility:

   Epidural physician approval
6. At the end of the birth fetal blood sample taken from the placenta for testing the level of paracetamol.
7. At the end of a blood sample taken birth for the client in liver function tests.
8. Interview woman with postpartum questionnaire will be made during her stay in the maternity ward.

Filling out a questionnaire that includes demographic data and about the process of birth, medical records.

ELIGIBILITY:
Inclusion Criteria:

* latent phase of labour
* low risk

Exclusion Criteria:

* high risk
* allergy to paracetamol
* liver insufficiency

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18+
Enrollment: 150 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-04-20 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
pain score | pain assessmant by vas scale during the latent phase of labor at delivery room. the data will be presented through study completion, an average of 1 year
  vas

SECONDARY OUTCOMES:
level of paracetamol | at the end of labor , blood samples from the mother and from the umbelical cord. the data will be presented through study completion, an average of 1 year
  samples of blood
pain experience | 72 hours after labor , the data will be presented through study completion, an average of 1 year
  pain scores by vas scale 0-10 scale. 0 no pain- 10 sever pain
pain influences | 72 hours after labor, the data will be presented through study completion, an average of 1 year
  influences of pain on daily activities, BPI scale behavioral pain scale , the inflouences of pain on movement, breast feeding, taking a bath, talking with visitors, 0- no influencs, 10 very much
pain experience and analgesia | 72 hours after labor, the data will be presented through study completion, an average of 1 year
  analgesia, which kind of analgesia medicines had used

IPD SHARING:
Plan to Share IPD: Undecided